CLINICAL TRIAL: NCT04549064
Title: Identification of AREG for the Detection of Pancreatic Cancer By Biosensor
Brief Title: Biomarkers of Pancreatic Cancer and New Way to Detection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: West China Hospital (Other); Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: 81672921
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum from pancreatic cancer patients and healthy controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with pancreatic cancer: Patients with pancreatic cancer did not receive any anti-cancer treatment and had no history of other malignant tumors.The diagnosis of pancreatic cancer patients is based on the final pathological diagnosis; the cancer staging is based on AJCC staging manual.
  Interventions: Diagnostic Test: diagnosis of pancreatic cancer
- Healthy Control: healthy controls had no history of benign pancreatic diseases and other benign and malignant tumors.
  Interventions: Diagnostic Test: diagnosis of pancreatic cancer

INTERVENTIONS:
Diagnostic Test: diagnosis of pancreatic cancer — Diagnosis of pancreatic cancer based on the concentration of serum biomarkers

SUMMARY:
Amphoteric regulatory protein (AREG), a member of epidermal growth factor (EGF) family, is expressed in many tumors.Our study confirmed that the expression of AREG in the serum of patients with pancreatic cancer is significantly higher than that of patients with benign pancreatic diseases and healthy people, which is expected to become a new early serum marker of pancreatic cancer. The serum concentration of AREG was detected by traditional ELISA and compared with CA-199, which was a conventional tumor marker of pancreatic cancer. Next, we compare the advantages of using sensor to detect AREG compared with ELISA.

DETAILED DESCRIPTION:
Serum was collected ： pancreatic cancer : healthy control =200:200 Clinical data were collected: age, gender, diagnosis, cancer stage, CA199 level at initial diagnosis, histopathological type, etc. The informed consent of the subjects was obtained before the study, and all experimental procedures were approved by ethics.

Draw a summary table of patient characteristics. The level of AREG was detected by ELISA kit and compared with CA199.

Fabrication of a new electrochemical biosensor. Characterization of sensor performance.

ELIGIBILITY:
Inclusion Criteria:

* The healthy control group had no history of benign pancreatic diseases and other benign and malignant tumors.
* Patients with pancreatic cancer did not receive any anti-cancer treatment and had no history of other malignant tumors.The diagnosis of pancreatic cancer patients is based on the final pathological diagnosis; the cancer staging is based on AJCC staging manual.

Exclusion Criteria:

* Uncontrolled active infection.
* Acute or chronic pancreatitis.
* It is accompanied by other uncontrolled malignant tumors.
* Any other uncontrolled active disease that prevents participation in the trial.
* Having a history of mental illness that is difficult to control.
* In the opinion of the investigator, the presence of medical or psychiatric history or laboratory abnormalities may increase the risk associated with participation in the study or the administration of the study drug, or may interfere with the interpretation of the results.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Total collection of pancreatic cancer: healthy control about 300：300. The study population met the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Pancreatic Cancer | through study completion, an average of 1 year
  Diagnosis based on the concentration of serum biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: han su xia, professor, Study Chair — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided